CLINICAL TRIAL: NCT04552145
Title: Physical Therapy Versus Surgical Decompression for Lumbar Spinal Stenosis: A Multicenter Randomized Controlled Trial
Brief Title: Physical Therapy vs Surgical Decompression for Lumbar Spinal Stenosis
Acronym: PTvsSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Sykehuset Innlandet HF (Other); Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/283
Record Dates: First submitted 2020-09-10; First posted 2020-09-17 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Spinal Stenosis
Keywords: Surgery; Physical Therapy Modalities
MeSH Terms: conditions — Spinal Stenosis | interventions — Surgical Procedures, Operative; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Randomised controlled multicenter study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgery (Active Comparator): Decompression surgery
  Interventions: Procedure: surgery
- physiotherapy (Active Comparator): Physical therapy program
  Interventions: Behavioral: Physiotherapy

INTERVENTIONS:
Procedure: surgery — standard decompression surgery
  Arms: surgery
Behavioral: Physiotherapy — 3 month physical therapy treatment including home activity based on a well defined program and 4 to 6 visits at physical therapy intervention center.
  Arms: physiotherapy

SUMMARY:
This is a randomized controlled multicenter trail comparing physical therapy to surgical decompression in patients with lumbar spinal stenosis. The 0-hypothesis is that there is no difference in the efficacy of structured physical therapy compared to surgical decompression.

Our aim is to evaluate if physical therapy can serve as a nonsurgical alternative for patients with LSS, where the severity of symptoms indicates the need of surgical decompression.

ELIGIBILITY:
Inclusion Criteria:

* Patients describing intermittent neurogenic claudication when walking and symptoms revealed by flexion of the spine.
* MRI shows lumbar spinal stenosis in one or two levels measured.
* The duration of the symptoms is longer than six months
* The patient is a candidate for surgical treatment
* The patient is capable of physical exercise

Exclusion Criteria:

* Vascular intermittent claudication
* Lumbar spinal stenosis in more than two levels
* Previous low back surgery
* Symptomatic lumbar disc herniation
* Degenerative scoliosis with Cobbs angle 30 degrees or more
* Degenerative spondylolisthesis grade 2 or more
* Spondylolysis with spondylolisthesis
* Recent osteoporotic fractures in the spine (last 6 month)
* Severe symptomatic arthrosis in hip or knee
* Locally advanced or metastatic cancer
* ASA >3
* Polyneuropathy recognized by neurography
* Insufficient Norwegian language skills

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
The proportion (%) of patients who improve 30% or more relative to baseline in Oswestry Disability Index 2.1 (ODI) | 6 months after index treatment
  Oswestry Disability Index 2.0 (ODI) is the most commonly used condition-specific outcome measure for spinal disorders in general. The score ranges from 0 to 100, with a lower score indicating less severe pain and disability. It has been validated into Norwegian and tested for psychometric properties.

SECONDARY OUTCOMES:
Patient reported leg pain by Numeric Rating Scale (NRS) | Baseline and 6 months
  NRS, scores 0-10, where a higher score indicates more pain
Patient reported leg pain by Numeric Rating Scale (NRS) | Baseline and 1 year
  NRS, scores 0-10, where a higher score indicates more pain
Patient reported leg pain by Numeric Rating Scale (NRS) | Baseline and 2 years
  NRS, scores 0-10, where a higher score indicates more pain
Patient reported back pain by Numeric Rating Scale (NRS) | Baseline and 6 months
  NRS, scores 0-10, where a higher score indicates more pain
Patient reported back pain by Numeric Rating Scale (NRS) | Baseline and 1 year
  NRS, scores 0-10, where a higher score indicates more pain
Patient reported back pain by Numeric Rating Scale (NRS) | Baseline and 2 years
  NRS, scores 0-10, where a higher score indicates more pain
Walking capacity measured by six-minutes walk-test | Baseline and 6 months
  Number of patients improving by 50 m or more after six-minutes walk-test
Improvement in health-related quality of life | Baseline and 1 year, and 2 years after index treatment
  Measured by EuroQol 5-dimensional 5-level questionnaire (EQ-5D-5L) utility index
Improvement in health-related quality of life | Baseline and 2 years
  Measured by EuroQol 5-dimensional 5-level questionnaire (EQ-5D-5L) utility index
Fraction of patients crossing over from physical therapy to surgical decompression | 6 months
  We will give the possibility to cross over to surgery 6 months, 1 year, and 2 years after index treatment
Fraction of patients crossing over from physical therapy to surgical decompression | 1 year
  We will give the possibility to cross over to surgery 6 months, 1 year, and 2 years after index treatment
Improvement of walking and standing capacity measured with accelerometer | Baseline and 6 months
  We will use a body-worn tri-axial lightweight accelerometer (AX3 sensor from Axivity, York, UK) attached by a waterproof tape to the midpoint of the patients' anterior right thigh and at the lower back.
  Daily physical activity such as walking, running, standing, sitting, lying down and cycling will be monitored. By comparing the continuous activity for one week before treatment, for one week at six-, and 12-month follow-up, we will be able to objectively report about changes in the activity level (25). Since LSS-patients have symptoms while walking and standing, we will report the activity as ratios of walking/standing compare to other activity, as well as summon the three longest walking/standing periods before and after treatment.
Improvement of walking and standing capacity measured with accelerometer | Baseline and 1 year
  We will use a body-worn tri-axial lightweight accelerometer (AX3 sensor from Axivity, York, UK) attached by a waterproof tape to the midpoint of the patients' anterior right thigh and at the lower back.
  Daily physical activity such as walking, running, standing, sitting, lying down and cycling will be monitored. By comparing the continuous activity for one week before treatment, for one week at six-, and 12-month follow-up, we will be able to objectively report about changes in the activity level (25). Since LSS-patients have symptoms while walking and standing, we will report the activity as ratios of walking/standing compare to other activity, as well as summon the three longest walking/standing periods before and after treatment.
The proportion (%) of patients who improve 30% or more relative to baseline in Oswestry Disability Index 2.1 (ODI) | 1 year after index treatment
  The ODI score ranges from 0 to 100, with a lower score indicating less severe pain and disability.
The proportion (%) of patients who improve 30% or more relative to baseline in Oswestry Disability Index 2.1 (ODI) | 2 years after index treatment
  The ODI score ranges from 0 to 100, with a lower score indicating less severe pain and disability.

CONTACTS AND LOCATIONS:
Overall Officials: Greger Lønne, md phd, Principal Investigator — Norwegian University of Science and Technology, Fac MH, INB; Jorunn L Helbostad, phd prof, Study Director — Norwegian University of Science and Technology, Fac MH, INB
Locations (3):
- Norway (3):
  - Innlandet Hospital Trust, Lillehammer
  - Martina Hansen's Hospital, Oslo
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No